CLINICAL TRIAL: NCT00556114
Title: A Pilot Study of Functional Optical Coherence Tomography for Ocular Imaging
Status: Completed | Type: Observational
Sponsor: University of California, Irvine (Other)
Collaborators: Beckman Laser Institute University of California Irvine (Other)
Responsible Party: Principal Investigator, Beckman Laser Institute and Medical Center, Baruch D. Kuppermann, M.D., Ph.D.,Professor Department of Ophthalmology and Biomedical Engineering, University of California, Irvine
Other Study IDs: 20043555
Record Dates: First submitted 2007-11-07; First posted 2007-11-09 (Estimated); Last update posted 2022-10-20 (Actual); Status verified 2022-10

CONDITIONS: Glaucoma; Diabetic Retinopathy; Age-Related Macular Degeneration; Central Retinal Vein Occlusion; Branch Retinal Vein Occlusion
Keywords: eye exam; Retina
MeSH Terms: conditions — Glaucoma; Diabetic Retinopathy; Macular Degeneration; Retinal Vein Occlusion | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Optical Coherence Tomography: Optical Coherence Tomography
  Interventions: Device: Optical Coherence Tomography

INTERVENTIONS:
Device: Optical Coherence Tomography — Optical Coherence Tomography

SUMMARY:
Growing evidence shows that altered blood flow plays a major role in many vision-threatening diseases including glaucoma, diabetic retinopathy, age-related macular degeneration, Central Retinal Vein Occlusion, and Branch Retinal Vein Occlusion. Optical coherence tomography, an established imaging technique use for eye exam in clinical ophthalmology, provides high-resolution cross sectional images of the retina and has increased our ability to understand many eye diseases.

DETAILED DESCRIPTION:
Optical Coherence Tomography is a non-invasive technique use a broadband light source to illuminate the area of study with light in the near infrared spectrum, then obtains static images of tissue structure from interference signals of the back-reflected light.

Optical Coherence Tomography a non-contact, non-invasive means of documenting both tissue structure and blood flow changes in ocular disease and can provide high resolution cross-sectional images of tissue structure, direct visualization of blood flow in blood vessels of the eye.

ELIGIBILITY:
Inclusion Criteria:

* Adult 18 years and older with normal eye, or has been diagnosed with eye disease.

Exclusion Criteria:

* Less than 18 years of age.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Primary care clinic and community sample.
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2007-01; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Medical exam tool | 24 hours
  Optical Coherence Tomography imaging technique of the retina and ability to diagnose and manage many eye diseases

CONTACTS AND LOCATIONS:
Overall Officials: Baruch D Kuppermann,, M.D., Ph.D., Principal Investigator — Ophthamology, University of California,Irvine; Zhongping Chen, Ph,D, Principal Investigator — Beckman Laser Institute University of California Irvine
Locations (1):
- Beckman Laser Institute, University of California,Irvine, Irvine, California, United States